CLINICAL TRIAL: NCT01983072
Title: Effect of Starter Formula With Symbiotic on Microbiota Balance
Brief Title: Symbiotic & Colonization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 06.08.INF
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: colonization of the gastrointestinal tract with bacteria
MeSH Terms: interventions — Infant Formula; Lactation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Infant starter formula (Active Comparator): standard infant formula
  Interventions: Dietary Supplement: Infant formula
- Infant starter formula + prebiotics + probiotics (Experimental): infant formula
  Interventions: Dietary Supplement: Infant formula
- Breastfeeding group (Other): reference group
  Interventions: Other: Breastfeeding

INTERVENTIONS:
Dietary Supplement: Infant formula
  Arms: Infant starter formula; Infant starter formula + prebiotics + probiotics
Other: Breastfeeding — Breastfeeding
  Arms: Breastfeeding group

SUMMARY:
The clinical trial aims at showing efficacy of prebiotics and the probiotic on microbiota balance. Together, the prebiotic solution in combination with the probiotic is expected to harmonize the microbiota of formula fed neonates with the microbiota of breast fed neonates and to allow a greater diversity of Bifidobacteria species in comparison with a formula non-supplemented with pre and probiotics.

DETAILED DESCRIPTION:
The infants will be recruited and randomized between 0 and 14 days. The intervention period, in terms of data necessary for the primary outcome, will be until they reach 3 months old. Measurements will be collected on three separate occasions during this period, i.e. 2 and 6 weeks and 3 months. Stools will be collected, on 3 separate occasions, i.e. 4-5 day, 6 weeks and 3 months of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infant
* Full term infant (≥ 37 weeks gestation; ≤ 42 weeks gestation)
* Age of infant is between 14 days at the time of enrollment
* Birth weight between 2500g and 4500g
* For the Formula fed groups: The infant's mother has elected, before the 14th day of their child's life, not to continue breastfeeding (no breastfeeding after the 14th day of the child's life) For the Breastfed group: The infant's mother has elected to fully breastfeed her baby, from enrollment to at least 3 months of age
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Congenital illness or malformation that may affect normal growth
* Significant pre-natal and/or post-natal disease
* Re-hospitalization for more than 2 days in the first 14 days of life. (Exceptionally, infants re-hospitalized because of jaundice may be enrolled in the study).
* Newborn who have received antibiotics during the first 14 days of life
* Receiving infant formula containing pro and/or prebiotics at the time of enrolment
* Newborn whose parents / caregivers cannot be expected to comply with treatment
* Newborn currently participating in another clinical trial

Max Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
stool bacterial populations | 3 months
  (Lactobacilli, Clostridia, Bacteroides, bifidobacteria, staphylococci, Enterobacteria and Bifidobacterial species at 1.5 months and 3 months of age of the infants.

SECONDARY OUTCOMES:
changes in weight | 3 months
  weight
Digestive tolerance (stool characteristics and frequency, vomiting, regurgitation, frequency of colic) | 3 months
  Digestive tolerance (stool characteristics and frequency, vomiting, regurgitation, frequency of colic)
changes in length | 3 months
  changes in length

CONTACTS AND LOCATIONS:
Overall Officials: Hania Szajewska, Principal Investigator — The Medical University of Warsaw
Locations (4):
- France (3):
  - Hôpital Saint Joseph, Marseille
  - Hôpital de la Conception, Marseille
  - Hôpital Nord, Marseille
- The Medical University of Warsaw, Warsaw, Poland